CLINICAL TRIAL: NCT06110585
Title: Transcranial Magnetic Stimulation: Evaluation of Improvement of Transdiagnostic Psychiatric Symptoms and Changes in Functional Neuroiming in Young Adults Patients With Major Depressive Disorder and Non-suicidal Self-injury
Brief Title: Transcranial Magnetic Stimulation in Patients With Depression and Non-suicidal Self-injury
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Brain Institute of Rio Grande do Sul (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 908; INSCER908 (Other: BrainInstitute)
Record Dates: First submitted 2023-10-11; First posted 2023-10-31 (Actual); Last update posted 2023-10-31 (Actual); Status verified 2023-10

CONDITIONS: Depressive Disorder, Major; Self-Injurious Behavior
MeSH Terms: conditions — Depressive Disorder, Major; Self-Injurious Behavior | interventions — Transcranial Magnetic Stimulation; salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: rTMS Treatment (Experimental): 20 sessions of TMS using the intermittent theta burst stimulation (iTBS) protocol
  Interventions: Procedure: Transcranial Magnetic Stimulation (TMS)
- Sham Comparator: Sham Treatment (Sham Comparator): 20 sham sessions using a placebo procedure with the TMS equipment.
  Interventions: Procedure: Sham

INTERVENTIONS:
Procedure: Transcranial Magnetic Stimulation (TMS) — The Intermittent Theta Burst Stimulation (iTBS) protocol will be used. This protocol involves bursts of stimulation at the theta frequency range, approximately 5 to 8 Hz. The specific combination utilized combines bursts of pulses at a frequency of 50 Hz, triggered at a rate of 5 Hz. Thus, a burst of 3 pulses is delivered with intervals of 20 ms between them, and this burst is repeated at intervals of 200 ms (i.e., 5 bursts per second). Every second, 15 pulses are delivered.
  Arms: Experimental: rTMS Treatment
Procedure: Sham — A stimulator with an arm containing a non-functional replica of the stimulation coil will be utilized. The application procedures will be identical to those of the active group, except that the device simulating the stimulation coil will not generate a magnetic field, only producing sound cues mimicking a stimulus.
  Arms: Sham Comparator: Sham Treatment

SUMMARY:
This clinical trial aims to investigate the effects of Transcranial Magnetic Stimulation (TMS) as an adjunctive treatment for young adult patients with depression and non-suicidal self-injury (NSSI).

The main questions this study aims to answer are:

* Does adjunctive TMS reduce psychiatric symptoms in young adults with major depressive disorder and non-suicidal self-injury?
* Does adjunctive TMS cause any changes in neuroimaging markers in young adults with major depressive disorder and non-suicidal self-injury?
* Does adjunctive TMS cause any effects on blood biomarkers in young adults with major depressive disorder and non-suicidal self-injury?

Participants in this study will undergo an extensive clinical evaluation, functional neuroimaging tests (MRI and fNIRS), and peripheral blood collection. They will be randomly assigned to one of two interventions: (1) 20 sessions of TMS using the intermittent theta burst stimulation (iTBS) protocol, or (2) 20 sham sessions using a placebo procedure with the TMS equipment. After the 20 sessions, additional clinical assessments, neuroimaging and blood tests will be conducted. The data analysis will compare the two groups in terms of response and remission of internalizing and externalizing psychiatric symptoms, as well as neuroimaging and blood tests outcomes.

DETAILED DESCRIPTION:
This comprehensive clinical trial seeks to explore the potential therapeutic benefits of Transcranial Magnetic Stimulation (TMS) when used as an adjunctive treatment for young adult patients grappling with both depression and non-suicidal self-injury (NSSI). The overarching objectives of this study are multifaceted and aim to address critical questions regarding the efficacy and underlying mechanisms of TMS in this particular demographic.

The primary research inquiries guiding this investigation are:

Psychiatric Symptom Reduction: Does the incorporation of adjunctive TMS lead to a significant reduction in psychiatric symptoms among young adults diagnosed with major depressive disorder and non-suicidal self-injury?

Neuroimaging Markers: Does adjunctive TMS induce any discernible changes in neuroimaging markers among young adults with major depressive disorder and non-suicidal self-injury? This involves employing sophisticated functional neuroimaging techniques such as MRI (Magnetic Resonance Imaging) and fNIRS (functional Near-Infrared Spectroscopy).

Blood Biomarkers: Are there observable effects on blood biomarkers in young adults with major depressive disorder and non-suicidal self-injury following adjunctive TMS treatment?

To investigate these questions, participants enrolled in the study will undergo an extensive and thorough clinical evaluation. Additionally, functional neuroimaging tests, encompassing both MRI and fNIRS, will be administered to gain insights into the neural correlates of TMS treatment. Furthermore, peripheral blood samples will be collected to analyze potential changes in blood biomarkers associated with TMS.

The study design incorporates a randomized assignment of participants to one of two interventions:

Active TMS Intervention: Participants will undergo 20 sessions of TMS utilizing the intermittent theta burst stimulation (iTBS) protocol.

Sham TMS Intervention: A control group will receive 20 sham sessions involving a placebo procedure with the TMS equipment.

Following the completion of the intervention phase, participants will undergo additional clinical assessments, neuroimaging, and blood tests to comprehensively evaluate the impact of TMS treatment. The subsequent data analysis will involve a rigorous comparison of the two groups, assessing factors such as the response and remission of internalizing and externalizing psychiatric symptoms, as well as outcomes related to neuroimaging and blood tests.

ELIGIBILITY:
Inclusion Criteria:

* Current diagnosis of major depressive disorder by the operational criteria of DSM-5 and non-suicidal self-injury behavior, defined by "engagement in and intentionally self-inflicted harm to the surface of one's body, likely resulting in bleeding, bruising, or pain (e.g., cutting, burning, puncturing, hitting, excessive rubbing), with the expectation that the injury will only lead to minor or moderate physical harm (i.e., no suicidal intent)". (at least one episode in the past year);
* Depression severity score ≥17 points (moderate depression criteria) on the 17-item Hamilton Depression Rating Scale (HAM-D-17);
* Currently receiving psychiatric treatment and/or engaged in psychotherapy with a minimum biweekly frequency;
* Consent to voluntary participation in the study, confirmed by signing the Informed Consent Form;
* Expressed willingness to comply with all study procedures, including imaging examinations and blood tests, with availability during the study, and to communicate with the study team regarding adverse events and other clinically important information;
* Commitment to access continuous psychiatric care before and after study completion;
* In good general health, as evidenced by medical history.

Exclusion Criteria:

* Participants who present pre-established contraindications for undergoing EMT, based on positive responses in the "TMS Adult Safety Screen (TASS)" questionnaire, such as: cochlear implants, brain stimulators (DBS), electrode implants or aneurysm clips, history of previous seizures, use of pacemakers, presence of implantable defibrillators, brain injury (whether vascular, neoplastic, traumatic, infectious, or metabolic);
* Patients who present a moderate to severe suicide risk, as determined by clinical evaluation or requiring psychiatric hospitalization during the recruitment or EMT application period;
* Patients with severe clinical comorbidities or any other reason that impedes self-mobility, preventing attendance at daily EMT sessions;
* Pregnant patients or those of childbearing age who are sexually active without using contraceptive methods.

Ages: 18 Years to 29 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-11-01 (Estimated); Primary Completion 2024-09-30 (Estimated); Study Completion 2025-02-28 (Estimated)

PRIMARY OUTCOMES:
Hamilton Depression Rating Scale | Week 1 prior to TMS treatment and week 1 after completion of TMS treatment
  Proportion of individuals with a 50% or more score reduction between before and after intervention
Patient Health Questionnaire-9 | Week 1 prior to TMS treatment and week 1 after completion of TMS treatment
  Proportion of individuals with a 50% or more score reduction between before and after intervention
Montgomery-Asberg Depression Rating Scale | Week 1 prior to TMS treatment and week 1 after completion of TMS treatment
  Proportion of individuals with a 50% or more score reduction between before and after intervention
fMRI assessed neural network connectivity | Week 1 prior to TMS treatment and week 1 after completion of TMS treatment
  Change on functional connectivity
fMRI-assessed resting connectivity | Week 1 prior to TMS treatment and week 1 after completion of TMS treatment
  Change (e.g. normalization) of baseline network-level deficits.

SECONDARY OUTCOMES:
Functional Assessment of Self-Mutilation (FASM) | Week 1 prior to TMS treatment and week 1 after completion of TMS treatment
  Difference in score between before and after the intervention
Hamilton Depression Rating Scale | 1, 3 , 6 and 12 months after completion of TMS treatment
  Proportion of individuals with a 50% or more score reduction between before and after intervention
Patient Health Questionnaire-9 | 1, 3 , 6 and 12 months after completion of TMS treatment
  Proportion of individuals with a 50% or more score reduction between before and after intervention
Montgomery-Asberg Depression Rating Scale | 1, 3 , 6 and 12 months after completion of TMS treatment
  Proportion of individuals with a 50% or more score reduction between before and after intervention
fNIRS- assessed changes in blood oxygenation levels in the brain | Week 1 prior to TMS treatment and week 1 after completion of TMS treatment
  Changes in blood oxygenation levels in the brain measured by fNIRS (functional near-infrared spectroscopy) to infer neural activity
Brain-Derived Neurotrophic Factor (BDNF) | Week 1 prior to TMS treatment and week 1 after completion of TMS treatment
  Changes in BDNF levels comparing pre- and post-treatment
Ciliary Neurotrophic Factor (CNTF) | Week 1 prior to TMS treatment and week 1 after completion of TMS treatment
  Changes in CNTF levels comparing pre- and post-treatment
Glial Cell-Derived Neurotrophic Factor (GDNF) | Week 1 prior to TMS treatment and week 1 after completion of TMS treatment
  Changes in GDNF levels comparing pre- and post-treatment
Nerve Growth Factor (NGF) | Week 1 prior to TMS treatment and week 1 after completion of TMS treatment
  Changes in GDNF levels comparing pre- and post-treatment

CONTACTS AND LOCATIONS:
Overall Officials: Lucas Spanemberg, PhD, Principal Investigator — Instituto do Cérebro do Rio Grande do Sul
Locations (1):
- Instituto do Cérebro do Rio Grande do Sul, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No